CLINICAL TRIAL: NCT05171907
Title: Application of Dietary Guidelines for the Brazilian Population by Teleconsultation for Patients With Obesity in Primary Health Care: A Randomized Clinical Trial
Brief Title: Application of Dietary Guidelines for the Brazilian Population by Teleconsultation in Obesity in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0128
Record Dates: First submitted 2021-07-29; First posted 2021-12-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Obesity
Keywords: Obesity; Chronic Disease; Noncommunicable Diseases; Telemedicine; Diet, Healthy; Primary Health Care; Unified Health System
MeSH Terms: conditions — Obesity; Chronic Disease; Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: A pragmatic multicentre randomised controlled trial, open-label, allocation at 1 : 1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients into the control group will receive the same assessments as patients in the intervention group, for the same time (in 1th, 8th, 24, and 48 weeks), but they will not receive nutritional teleconsultation.
- Intervention Group (Other): Teleintervention based on Dietary Guidelines for the Brazilian Population during 8 weeks; two subsequent assessments will also be made, in 24th and 48th weeks, to assess the maintenance of weight loss.
  Interventions: Behavioral: Teleobesity

INTERVENTIONS:
Behavioral: Teleobesity — Teleintervention based on Dietary Guidelines for the Brazilian Population during 8 weeks; two subsequent assessments will also be made, in 24th and 48th weeks, to assess the maintenance of weight loss.
  Arms: Intervention Group

SUMMARY:
Obesity is a chronic disease that is highly prevalent in Brazil. It is associated with diabetes and hypertension. Obesity may decrease quality of life. Communication tools, such as mobile devices and social media, are helping to control and prevent obesity. In this 2-arm randomized clinical trial, the investigators aim to evaluate the efficacy of the Dietary Guidelines for the Brazilian Population through 8 weekly video nutritional monitoring sessions with nutritionists. Both groups will receive guidance from reference professionals from primary health care (physician and nurse). Throughout the intervention program, both groups will be equally evaluated in order to verify at the end of the study effectiveness in weight loss and life quality improvement.

DETAILED DESCRIPTION:
Obesity is a multifactorial disease of epidemic proportions worldwide. The use of telecommunication tools has been used in health and nutrition in different contexts, seeking to reduce the burden of non-communicable chronic diseases. Telehealth interventions are effective to increase quality of life and to improve the dietary food intake of participants; this kind of treatment seems feasable, cost-effective and has promising results to induce weight loss in obese individuals. This project will evaluate the impact of a remote nutritional intervention in short (8 weeks) and long term (24 and 48 weeks) on the weight fo obese individuals. The intervention will be based on the Dietary Guidelines for the Brazilian Population. It will focus on primary care patients and will have a multidisciplinary approach. It is an open-label pragmatic multicentre randomized controlled trial, with an 1:1 allocation: (1) intervention group (n = 289): Remote consultation with nutritionists based on the Dietary Guidelines for the Brazilian Population; (2) control group (n = 289): usual follow-up in Primary Health Care (PHC). The primary outcome will be weight change at 8 weeks. Additionally, the investigators will evaluate food consumption and quality of life at 8 and 24 weeks as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female and male individuals, with BMI ≥30 kg/m²;
* Age over 18 years;
* Internet access by phone or tablet or computer and WhatsApp multi-platform application (Facebook Inc.);
* Weekly time availability (10-20 minutes).

Exclusion Criteria:

* Individuals who do not have access to the WhatsApp multi-platform application (Facebook Inc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 578 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-22 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Weight change | 8 weeks
  Weight change, measured using a calibrated scale at a Primary Health Care health unit, at the end of 8 weeks.

SECONDARY OUTCOMES:
Food consumption improvement | 8 and 24 weeks
  Improvement in food consumption measured through 24-hour dietary recall (R24h), at the end of 8th and 24th week.
Quality of life measured using the Short Form Health Survey 36 | 8 and 24 weeks
  Quality of life improvement measured using the Short Form Health Survey 36, SF-36, at the end of 8th and 24th week. The SF-36 presents a final score from 0 to 100, in which zero corresponds to the worst general health status and 100 the best health status.
Weight change (follow up) | 24 and 48 weeks
  Weight change, measured using a calibrated scale at a Primary Health Care health unit, at the end of 24 and 48 weeks of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Rodrigues Gonçalves, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil